CLINICAL TRIAL: NCT05403957
Title: A Cluster Randomised Controlled Trial on Tobacco Industry Denormalisation
Brief Title: A Cluster RCT on TID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Principle investigator and associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TIDvideo202021
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Tobacco Industry; Denormalisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TID video (Experimental)
  Interventions: Other: TID video
- TID worksheet (Active Comparator)
  Interventions: Other: TID worksheet
- SSB worksheet (Placebo Comparator)
  Interventions: Other: SSB worksheet

INTERVENTIONS:
Other: TID video — Main intervention: A video introducing the tobacco industry's marketing tactics to attract children and adolescents to smoke and their manipulation of tobacco control policy formation.
  Booster intervention: 6 screenshots from the video and 6 true or false questions.
  Arms: TID video
Other: TID worksheet — Main intervention: A worksheet using pictures and texts to introduce the tobacco industry's marketing tactics to attract children and adolescents to smoke and their manipulation of tobacco control policy formation.
  Booster intervention: 8 pictures from the TID worksheet in the main intervention and 6 true or false questions.
  Arms: TID worksheet
Other: SSB worksheet — Main intervention: A worksheet using pictures and texts to introduce the beverage industry's marketing tactics to attract children and adolescents to drink SSBs and the health risks of SSBs.
  Booster intervention: 8 pictures from the SSB worksheet in the main intervention and 6 true or false questions.
  Arms: SSB worksheet

SUMMARY:
The brief intervention comprised the main intervention (tobacco industry denormalisation [TID] video, TID worksheet and sugar-sweetened beverages [SSB] worksheet) and booster intervention (worksheets where key contents in the main intervention reappeared).

The worksheets in the main intervention were printed in colour and contained eight pictures and eight texts which described the pictures. Students needed to match the pictures and texts. The booster worksheets contained the previous eight coloured pictures for the TID and SSB worksheet groups or six coloured screenshots from the TID video. Students needed to complete the six true or false questions based on the pictures provided.

Assessments were conducted immediately (T1), two weeks (T2), one month (T3) and three months (T4) after the main intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents' consent to their children's participation;
* Parents and children could understand Chinese.

Exclusion Criteria:

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2881 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
TID beliefs | Immediately after the main intervention
  1. Tobacco industry's philanthropy is to care about community well-being.
  2. Tobacco industry does everything possible to make children smoke.
  3. Tobacco industry deceives the public for commercial gain.
  4. Tobacco industry uses many tactics to resist tobacco control regulations.
  All the statements have 5 options from strongly disagree to strongly agree. The options were scored as 1-5 or 5-1, as appropriate, with higher scores indicating stronger TID beliefs.
Alternative smoking product (ASP)-related knowledge | Immediately after the main intervention
  Electronic cigarettes (ECs) and heated tobacco products (HTPs) are less harmful than cigarettes.
  The statement has 5 options from strongly disagree to strongly agree. The options were scored as 5-1, with higher scores indicating better knowledge.
Risk perceptions of ASPs | Immediately after the main intervention
  1. Do you think trying a few puffs of ECs will harm your health?
  2. Do you think trying a few puffs of HTPs will harm your health?
  Both statements have 11 options from not harmful at all to very harmful. The options were scored as 0-10, with higher scores indicating stronger anti-tobacco attitudes.
Acceptability of ASPs | Immediately after the main intervention
  1. Do you think it is acceptable for primary school students to try a few puffs of ECs?
  2. Do you think it is acceptable for primary school students to try a few puffs of HTPs?
  Both statements have 11 options from very unacceptable to very acceptable. The options were scored as 0-10, with lower scores indicating stronger anti-tobacco attitudes.
General views on the tobacco industry | Immediately after the main intervention
  What do you think of the tobacco industry?
  The statement has 11 options from very bad to very good. The options were scored as 0-10, with lower scores indicating stronger anti-tobacco attitudes.

SECONDARY OUTCOMES:
Susceptibility to use ASPs | Immediately after the main intervention
  1. If your good friend passes you an EC, will you use it?
  2. Do you think you will use EC within the next 12 months?
  3. If your good friend passes you an HTP, will you use it?
  4. Do you think you will use HTP within the next 12 months?
  All the statements have 5 options from definitely yes to definitely not. Responses were dichotomised as a binary outcome, students who chose "definitely not" for both items were deemed not susceptible to a specific smoking product and otherwise susceptible.
TID beliefs | One month after the main intervention
  1. Tobacco industry conceals the harms of smoking products for commercial gain.
  2. Tobacco industry deceives the public for commercial gain.
  3. Tobacco industry uses many tactics to resist tobacco control regulations.
  All the statements have 5 options from strongly disagree to strongly agree. The options were scored as 1-5, with higher scores indicating stronger TID beliefs.
ASP-related knowledge | One month after the main intervention
  1. ECs and HTPs are less harmful than cigarettes.
  2. HTPs contain many carcinogens.
  Both statements have 5 options from strongly disagree to strongly agree. The options were scored as 1-5 or 5-1, as appropriate, with higher scores indicating better knowledge.
Risk perceptions of ASPs | One month after the main intervention
  1. Do you think trying a few puffs of ECs will harm your health?
  2. Do you think trying a few puffs of HTPs will harm your health?
  Both statements have 11 options from not harmful at all to very harmful. The options were scored as 0-10, with higher scores indicating stronger anti-tobacco attitudes.
Acceptability of ASPs | One month after the main intervention
  1. Do you think it is acceptable for primary school students to try a few puffs of ECs?
  2. Do you think it is acceptable for primary school students to try a few puffs of HTPs?
  Both statements have 11 options from very unacceptable to very acceptable. The options were scored as 0-10, with lower scores indicating stronger anti-tobacco attitudes.
General views on the tobacco industry | One month after the main intervention
  What do you think of the tobacco industry?
  The statement has 11 options from very bad to very good. The options were scored as 0-10, with lower scores indicating stronger anti-tobacco attitudes.
Susceptibility to use ASPs | One month after the main intervention
  1. If your good friend passes you an EC, will you use it?
  2. Do you think you will use EC within the next 12 months?
  3. If your good friend passes you an HTP, will you use it?
  4. Do you think you will use HTP within the next 12 months?
  All the statements have 5 options from definitely yes to definitely not. Responses were dichotomised as a binary outcome, students who chose "definitely not" for both items were deemed not susceptible to a specific smoking product and otherwise susceptible.
TID beliefs | Three months after the main intervention
  1. Tobacco industry uses many tactics to resist tobacco control regulations.
  2. Tobacco industry struggles to build a corporate image to improve tobacco products sales.
  Both statements have 5 options from strongly disagree to strongly agree. The options were scored as 1-5, with higher scores indicating stronger TID beliefs.
ASP-related Knowledge | Three months after the main intervention
  1. HTPs contain many carcinogens.
  2. ECs are less harmful than cigarettes.
  3. Secondhand aerosols of ECs and HTPs are less harmful.
  All the statements have 5 options from strongly disagree to strongly agree. The options were scored as 1-5 or 5-1, as appropriate, with higher scores indicating better knowledge.
Risk perceptions of ASPs | Three months after the main intervention
  1. Do you think trying a few puffs of ECs will harm your health?
  2. Do you think trying a few puffs of HTPs will harm your health?
  Both statements have 11 options from not harmful at all to very harmful. The options were scored as 0-10, with higher scores indicating stronger anti-tobacco attitudes.
Acceptability of ASPs | Three months after the main intervention
  1. Do you think it is acceptable for primary school students to try a few puffs of ECs?
  2. Do you think it is acceptable for primary school students to try a few puffs of HTPs?
  Both statements have 11 options from very unacceptable to very acceptable. The options were scored as 0-10, with lower scores indicating stronger anti-tobacco attitudes.
General views on the tobacco industry | Three months after the main intervention
  What do you think of the tobacco industry?
  The statement has 11 options from very bad to very good. The options were scored as 0-10, with lower scores indicating stronger anti-tobacco attitudes.
Susceptibility to use ASPs | Three months after the main intervention
  1. If your good friend passes you an EC, will you use it?
  2. Do you think you will use EC within the next 12 months?
  3. If your good friend passes you an HTP, will you use it?
  4. Do you think you will use HTP within the next 12 months?
  All the statements have 5 options from definitely yes to definitely not. Responses were dichotomised as a binary outcome, students who chose "definitely not" for both items were deemed not susceptible to a specific smoking product and otherwise susceptible.

CONTACTS AND LOCATIONS:
Overall Officials: SAI YIN HO, Principal Investigator — The University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No